CLINICAL TRIAL: NCT07255885
Title: CRYSTALSIGHT: ''Cohort 1.5" Clinical Investigation Study With OCCUTRACK and Tan Tock Seng Eye Clinic to Further Develop Remote Monitoring of Maculopathy at Home Using Artificial Intelligence for Eye Tracking
Status: Completed | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Occutrack Medical Solutions Pte Ltd (Unknown); Agency for Science, Technology and Research (Other); National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Laude Augustinus, Senior Consultant, Tan Tock Seng Hospital
Other Study IDs: 2024-3478
Record Dates: First submitted 2025-03-17; First posted 2025-12-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Maculopathy; Maculopathy, Age Related; Macular Degeneration, Age-Related; Diabetic Retinopathy; Wet Age Related Macular Degeneration; Aged-related Macular Degeneration
Keywords: gaze-tracking
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRYSTALSIGHT: Presenting stimulus targets while using Crystalsight: The test presents three types of targets and assesses corresponding gaze responses in pseudorandom succession on the screen. During this, the Crystalsight AI uses a high-definition camera to perform eye-gaze tracking to generate data coordinates of eye movement.
  Interventions: Device: CRYSTALSIGHT Test

INTERVENTIONS:
Device: CRYSTALSIGHT Test — Eye gaze tracking tests will be automated, and patients will only need to follow through with the stimulus/image shown without physical contact with the eye gaze tracker using CRYSTALSIGHT and Tobii. A series of stimulus dots in the form of a pursuit (moving stimulus) or saccade (fixed stimulus and fixed speed) will be presented on the screen and the user under test (UAT) will need to look at the targets presented. The test is similar to Microperimetry and Humphrey's visual field test. A score will be generated at the end of the test.
  Research Procedure:
  1. CRYSTALSIGHT
  2. Tobii
  Subjects perform the CRYSTALSIGHT test monocularly and pursue a pre-determined target moving in a customized waveform across the computer screen. The trail of the gaze points generated by the subject following the target is simultaneously recorded and stored.
  Eye dilation will not be required for the purpose of this research study as fundoscopy nor OCT imaging will not be performed.

SUMMARY:
The development of a next-generation 'CRYSTALSIGHT' solution using combinations of a novel and cost-effective eye-tracking system with artificial intelligence-based eye-tracking algorithms that detect macular abnormalities and enable clinicians to review and monitor the prognosis of patients via a web platform through the following deliverables.

1. Evaluate and improve a home-monitoring regimen involving the self-tests of the CRYSTALSIGHT gaze-tracking system
2. To demonstrate that CRYSTALSIGHT has the same or superior gaze-tracking capacities as Tobii.
3. Evaluate the CRYSTALSIGHT device for its functionality and ease of use as a qualitative measurement tool for patients.
4. Develop the Design History File (DHF) for regulatory filing requirements.

   2. This study will improve on the existing gaze-based scoring methodology for disease activity monitoring over time (delta-change) by quantitatively measuring saccadic speed, pursuit and micro-saccades.

DETAILED DESCRIPTION:
Macula degeneration is more prevalent with ageing and can result in blurred or distorted vision, often accompanied by a dark patch blocking the center of the visual field. In the management of age-related macular degeneration (AMD), patients are required to attend regular check-ups at the specialist eye clinic by the clinician to monitor if their disease. The eye examinations that patients undergo during these clinic visits which may include fundoscopy and optical coherence tomography. A preventive treatment for exudative or wet AMD is the administration of an intravitreal injection of an anti-vascular endothelial growth factor (anti-VEGF) at these regular clinic sessions.

Although anti-vascular endothelial growth factor (VEGF) injections are an effective treatment for many patients with Wet-AMD, there are several unmet needs in treatment of AMD and none of them cures the disease or reverses its course. Some patients do not respond to VEGF injections. There are no standardized treatment schedules, there is a large treatment burden, and visual loss continues over time.

Additionally, the main drawback of anti-VEGF therapy is its high cost, which suppose a significant burden on health systems, and often makes such a regimen unaffordable in clinical practice. There is no treatment for GA. Therefore, the prevention of advanced disease like Wet-AMD and finding new and effective treatments remain a significant challenge. Advances in imaging and genetics and molecular technologies have led to the identification of new risk factors for disease progression, but not all have been evaluated in comprehensive prediction models. Perhaps, comprehensive prediction models could lead to the development of tailored, individualized therapy and improve the personalised healthcare.

As such, the application of this next-generation OCCUTRACK Technology to develop a comprehensive risk score algorithm and to estimate the risk scores to identify individuals at high risk for disease progression to advanced stages would result in earlier intervention and reduced burden of visual loss due to AMD. This approach could enable the tailored individualized Anti-VEGF Therapy to promote personalized medicine and improve the quality of life of patients with Wet-AMD.

A Proof-of-Concept (POC) was completed by TTSH clinician and AStar-I2R scientist to co-develop and patent a software - Automated Vision Assessment and Impairment Detection through Gaze Analysis (AVIGA). AVIGA is now referred to as "CRYSTALSIGHT" as part of the commercialization branding. A local medical incubator, Trendlines Medical Singapore, has licensed it from the research party. This led to the spin-off of a new company - Occutrack Pte Ltd to continue the collaboration with TTSH, focusing on the commercialization of the CRYSTALSIGHT. AVIGA previously used a costly commercial tobii gaze tracker that could potentially limit consumer adoption, the CRYSTALSIGHT system was designed to mitigate costs by incorporating an AI-augmented video camera with gaze tracking algorithms designed to provide a comprehensive assessment of a patient's vision. With this non-invasive technology, retinal specialists can monitor the real time progression and prognosis of patients with AMD while they are in the comfort of their own home without the need for manual or skilled intervention and expensive equipment.

This project proposal is to evaluate the performance and accuracy of the CRYSTALSIGHT technology as a tool for determining macular disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between ages 21 and 100
2. Both genders
3. Subjects with maculopathies
4. Ability to comply with the study protocol, in the investigator's judgment
5. Subjects must have the cognitive capacity to provide personal consent (i.e. no cognitively impaired persons will be recruited).

Exclusion Criteria:

1. Uncontrolled blood pressure, defined as systolic blood pressure >180 millimeters of mercury (mmHg) and/or diastolic blood pressure >100 mmHg while a patient is at rest.
2. Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study.
3. History of idiopathic or autoimmune-associated uveitis in either eye.
4. Active ocular inflammation or suspected or active ocular or periocular infection in either eye.
5. Other protocol-specified exclusion criteria may apply.
6. Individuals with indications of cognitive impairment and unable to make decisions for themselves to provide informed consent will be excluded from the study.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals will be voluntarily recruited from Tan Tock Seng Hospital (TTSH) Ophthalmology Specialist Outpatient Clinics after they have been assessed for eligibility based on established clinical diagnosis from the case notes through TTSH NGEMR. Informed consent will be obtained for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Agreement of CRYSTALSIGHT with Tobii Gaze Tracker for Macular Disease Monitoring | Baseline
  To assess the agreement between the CRYSTALSIGHT device and the commercial Tobii eye tracker in quantifying gaze parameters (e.g., saccadic velocity, pursuit stability, micro-saccades) in patients with maculopathies.

SECONDARY OUTCOMES:
Agnostic Concordance of CRYSTALSIGHT with Clinical Disease Activity | Baseline
  To assess whether CRYSTALSIGHT-generated scores correspond with disease activity levels as determined by standard clinical evaluations (e.g., OCT imaging, clinical diagnosis).
Rate of Incomplete or Failed Tests Using CRYSTALSIGHT | Baseline
  To determine the operational reliability of CRYSTALSIGHT by measuring the frequency of unsuccessful or incomplete tests due to user or device limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Augustinus Laude, MBChB, Principal Investigator — Tan Tock Seng Hospital; Zheng Kuang Noel Soh, BSc, Study Director — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawasaki R, Wang JJ, Aung T, Tan DT, Mitchell P, Sandar M, Saw SM, Wong TY; Singapore Malay Eye Study Group. Prevalence of age-related macular degeneration in a Malay population: the Singapore Malay Eye Study. Ophthalmology. 2008 Oct;115(10):1735-41. doi: 10.1016/j.ophtha.2008.02.012. Epub 2008 Apr 25. PMID 18439679
- [Background] Trevino R, Kynn MG. Macular function surveillance revisited. Optometry. 2008 Jul;79(7):397-403. doi: 10.1016/j.optm.2007.09.017. PMID 18577497
- [Background] Ai Ping Yow, Damon Wong, Huiying Liu, Hongyuan Zhu, Ivy Jing-Wen Ong, Laude A, Tock Han Lim. Automatic visual impairment detection system for age-related eye diseases through gaze analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:2450-2453. doi: 10.1109/EMBC.2017.8037352. PMID 29060394
- [Background] Mathew R, Sivaprasad S. Environmental Amsler test as a monitoring tool for retreatment with ranibizumab for neovascular age-related macular degeneration. Eye (Lond). 2012 Mar;26(3):389-93. doi: 10.1038/eye.2011.326. Epub 2011 Dec 16. PMID 22173073
- [Background] AREDS2-HOME Study Research Group; Chew EY, Clemons TE, Bressler SB, Elman MJ, Danis RP, Domalpally A, Heier JS, Kim JE, Garfinkel R. Randomized trial of a home monitoring system for early detection of choroidal neovascularization home monitoring of the Eye (HOME) study. Ophthalmology. 2014 Feb;121(2):535-44. doi: 10.1016/j.ophtha.2013.10.027. Epub 2013 Nov 8. PMID 24211172
- [Background] AREDS2 Research Group; Chew EY, Clemons T, SanGiovanni JP, Danis R, Domalpally A, McBee W, Sperduto R, Ferris FL. The Age-Related Eye Disease Study 2 (AREDS2): study design and baseline characteristics (AREDS2 report number 1). Ophthalmology. 2012 Nov;119(11):2282-9. doi: 10.1016/j.ophtha.2012.05.027. Epub 2012 Jul 26. PMID 22840421
- [Background] Chew EY, Clemons TE, Agron E, Sperduto RD, Sangiovanni JP, Davis MD, Ferris FL 3rd; Age-Related Eye Disease Study Research Group. Ten-year follow-up of age-related macular degeneration in the age-related eye disease study: AREDS report no. 36. JAMA Ophthalmol. 2014 Mar;132(3):272-7. doi: 10.1001/jamaophthalmol.2013.6636. PMID 24385141
- [Background] Age-Related Eye Disease Study Research Group. The Age-Related Eye Disease Study (AREDS): design implications. AREDS report no. 1. Control Clin Trials. 1999 Dec;20(6):573-600. doi: 10.1016/s0197-2456(99)00031-8. PMID 10588299
- [Background] Goldberg, J.H. and A.M. Wichansky, Eye tracking in usability evaluation: A practitioner's guide, in the Mind's Eye. 2003, Elsevier. p. 493-51
- [Background] Goldberg, J.H. and X.P. Kotval, Computer interface evaluation using eye movements: methods and constructs. International journal of industrial ergonomics, 1999. 24(6): p. 631
- [Background] Huiying Liu, Yanwu Xu, Damon Wong, Ai Ping Yow, Laude A, Tock Han Lim. Detecting impaired vision caused by AMD from gaze data. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:3142-3145. doi: 10.1109/EMBC.2017.8037523. PMID 29060564
- [Background] Huiying Liu, Wong D, Ai Ping Yow, Yanwu Xu, Fengshou Yin, Laude A, Tock Han Lim. Determining the difference in eyegaze measurements in individuals with age related macular degeneration. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:1348-1351. doi: 10.1109/EMBC.2016.7590957. PMID 28268575

DOCUMENTS (1):
  • Study Protocol (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT07255885/Prot_000.pdf